CLINICAL TRIAL: NCT03211195
Title: Bioequivalence Study Comparing Sotagliflozin Tablet Commercial Formulation (Test) and Sotagliflozin Tablet Development Formulation (Reference) in Healthy Male and Female Subjects Under Fasted Conditions
Brief Title: Sotagliflozin Bioequivalence Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BEQ15271; U1111-1197-7610 (Other: UTN)
Record Dates: First submitted 2017-07-06; First posted 2017-07-07 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sotagliflozin - Commerical (Experimental): Healthy volunteers will be administered a single dose Sotagliflozin (SAR439954) tablet (Commercial formulation) by mouth under fasted conditions
  Interventions: Drug: Sotagliflozin (SAR439954)
- Sotagliflozin -Development (Active Comparator): Healthy volunteers will be administered a single dose Sotagliflozin (SAR439954) tablet (Development formulation) by mouth under fasted conditions - Type: Active Comparator
  Interventions: Drug: Sotagliflozin (SAR439954)

INTERVENTIONS:
Drug: Sotagliflozin (SAR439954) — Pharmaceutical form: tablet
  Route of administration: oral

SUMMARY:
Primary Objective:

To determine the bioequivalence of a single dose of the commercial tablet of sotagliflozin (test) compared to the development tablet of sotagliflozin (reference) under fasting conditions in healthy male and female subjects.

Secondary Objectives:

* To evaluate the single-dose pharmacokinetics of sotagliflozin and its main metabolite sotagliflozin 3-O-glucuronide following administration of a single sotagliflozin (test) tablet or a single sotagliflozin (reference) table in healthy male and female subjects under fasting conditions.
* To evaluate safety and tolerability of a single dose sotagliflozin (test) tablet compared to a single sotagliflozin (reference) tablet administered under fasted conditions in healthy male and female subjects.

DETAILED DESCRIPTION:
The study duration per subject will be 36-99 days and will consist of a screening period of 2 to 21 days, a study period of 7 days for each of four periods, and a washout of 8-21 days between each dose administration, and a final follow up visit 10-15 days after final dose administration.

ELIGIBILITY:
Inclusion criteria :

* Healthy male and female subjects 18-55 years old inclusive, male or female.
* Certified as healthy by comprehensive clinical assessment (detailed medical history and complete physical examination).
* Body weight between 50.0 and 100.0 kg, inclusive if male, and between 40.0 and 90.0 kg, inclusive if female, Body mass index (BMI) of 18.0 to 30.0 kg/m2 inclusive.
* Normal vital signs, ECG and laboratory parameters.
* Female subjects must use a double contraception method including a highly effective method of contraception except if she has undergone sterilization at least 3 months earlier or is post-menopausal. Hormonal contraception is permitted in this study.
* Having given written informed consent prior to undertaking of study procedure.
* Covered by a health insurance system where applicable, and/or in compliance with the recommendation of the national laws in force relating to biomedical research.
* Not under any administrative or legal supervision.
* Male subjects, whose partners are of childbearing potential (including lactating women) must accept to use, during sexual intercourse, a double contraception method from the inclusion up to 3 months after the last dosing.
* Male subjects, who partners are pregnant, must use during sexual intercourse a condom from inclusion to three months after the last dosing.
* Male subject has agreed not to donate sperm from the time of inclusion up to 3 months after the last dosing.

Exclusion criteria:

* Any history or presence of clinically relevant disease at screening which could interfere with the objectives of the study or the safety fo the subject's participation.
* History of renal disease, or significantly abnormal kidney function test (glomerular filtration rate [GFR]<90 mg/min as calculated using the Cockcroft-Gault equation) at screening.
* Frequent headaches and/or migraines, recurrent nausea and/or vomiting.
* Blood donation of a pint or more within 2 months before inclusion.
* Symptomatic, postural hypotension, irrespective of the decrease in blood pressure, or asymptomatic postural hypotension defined as a decrease in systolic blood pressure of 20 mmHg or more within 3 minutes when changing from supine to standing position.
* Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician.
* Any history of presence of deep vein thrombosis or pulmonary embolism or a recurrent or frequent history of deep vein thrombosis in first degree relatives (parents, siblings, or children).
* Any presence or history of urinary tract infection or genital mycotic infection in the last 4 weeks before screening.
* History or presence of drug or alcohol abuse.
* Smoking more than 5 cigarettes or equivalent per day, unable to stop smoking during the study.
* Excessive consumption of beverages containing xanthine bases (more than 4 cups or glasses per day).
* If female, pregnancy (defined as positive beta-HCG) blood test if applicable) breast-feeding.
* Any medication (including St John's Wort) within 14 days before inclusion or within 5 time the elimination half-life or pharmacodynamic half-life of the medication; any vaccination within the last 28 days and any biologics (antibody or its derivatives) given within 4 months before inclusion or within 5 terminal elimination half-life of the biologic.
* Any subject in the exclusion period of a previous study according to applicable regulations.
* Any subject who cannot be contracted in the case of an emergency.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2017-08-22 (Actual); Study Completion 2017-08-22 (Actual)

PRIMARY OUTCOMES:
Assessment of PK (pharmacokinetic) parameter: Cmax | From 0 to 120 hours after SAR439954 intake
  Sotagliflozin: Maximum plasma concentration (Cmax)
Assessment of PK parameter: AUClast | From 0 to 120 hours after SAR439954 intake
  Sotagliflozin: Area under the concentration-time curve from 0 to last quantifiable concentration (AUClast)
Assessment of PK parameter: AUC | From 0 to 120 hours after SAR439954 intake
  Sotagliflozin: Area under the concentration-time curve from 0 to infinity

SECONDARY OUTCOMES:
Assessment of PK parameter: Tmax | From 0 to 120 hours after SAR439954 intake
  Sotagliflozin: Time to reach maximum plasma concentration (Tmax)
Assessment of PK parameter: t1/2 | From 0 to 120 hours after SAR439954 intake
  Sotagliflozin: Terminal elimination half life (T1/2)
Assessment of PK parameter: Vz/F | From 0 to 120 hours after SAR439954 intake
  Sotagliflozin: Apparent volume of distribution during terminal phase after non-intravenous administration Vz/F
Assessment of PK parameter: CL/F | From 0 to 120 hours after SAR439954 intake
  Sotagliflozin: Apparent total body clearance of a drug from the plasma (CL/F)
Assessment of PK parameter: Cmax | From 0 to 120 hours after SAR439954 intake
  Sotagliflozin 3-O-glucuronide: Maximum plasma concentration (Cmax)
Assessment of PK parameter: AUC | From 0 to 120 hours after SAR439954 intake
  Sotagliflozin 3-O-glucuronide: Area under the concentration-time curve from 0 to infinity
Assessment of PK parameter: AUClast | From 0 to 120 hours after SAR439954 intake
  Sotagliflozin 3-O-glucuronide: Area under the concentration-time curve from 0 to last quantifiable concentration (AUClast)
Assessment of PK parameter: Tmax | From 0 to 120 hours after SAR439954 intake
  Sotagliflozin 3-O-glucuronide: Time to reach maximum plasma concentration (Cmax)
Assessment of PK parameter: t1/2 | From 0 to 120 hours after SAR439954 intake
  Sotagliflozin 3-O-glucuronide: Terminal elimination half life (T1/2)
Treatment emergent adverse events (TEAE) | From 0 to 144 hours after SAR439954 intake
  Number treatment emergent adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 840001, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org